CLINICAL TRIAL: NCT04565925
Title: Sildenafil for Treatment of Urinary Incontinence in Patients With Spinal Cord Injuries
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-0197
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injuries; Urinary Incontinence
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Incontinence | interventions — Sildenafil Citrate; Lactose

STUDY DESIGN:
Intervention Model Description: Each subject will be administered both sildenafil 20mg TID for 4 weeks and placebo (lactose) TID for 4 weeks in a crossover fashion with a 2 week washout period between treatments.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Both the subjects and the investigators will be blinded to the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sildenafil 20mg TID then Placebo TID (Experimental): Subjects will be administered Sildenafil 20mg TID for 4 weeks. There will be a 2 week washout period then subjects will be administered Placebo (lactose) TID for 4 weeks.
  Interventions: Drug: Sildenafil Citrate; Drug: Placebo
- Placebo TID then Sildenafil 20mg TID (Experimental): Subjects will be administered Placebo (lactose) TID for 4 week. There will be a 2 week washout period and then subjects will be administered Sildenafil 20mg TID for 4 weeks.
  Interventions: Drug: Sildenafil Citrate; Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil Citrate — Sildenafil 20mg TID for 4 weeks
  Other Names: Revatio
Drug: Placebo — Placebo (Lactose) TID for 4 weeks
  Other Names: Lactose

SUMMARY:
The goal of this study is to determine whether administration of sildenafil will decrease urine leakage in patients with spinal cord injuries.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) is a devastating condition affecting 291,000 women and men in the US alone. Urinary incontinence (UI) is a common problem in these patients, affecting 52% of the population, with episodes of incontinence occurring daily in 20-27% of affected persons. UI after spinal cord injury (SCI) is a major cause of distress and morbidity amongst patients with SCI, and is associated with decreased quality of life in general, physical, and emotional domains. UI has the undesirable side effects of perineal irritation and infection, increased odor, disrupted sleep, embarrassment, need to change clothes/bedding, and sexual dysfunction, as well as significant financial burden. Persons living with a SCI have ranked urinary problems as the most important health problem after injury. Addressing this significant problem and providing relief has the potential to significantly improve the lives of patients with SCI.

Typical treatment options are geared toward the type of UI in each patient. For stress UI, the goal of treatment is to provide support to the pelvic floor and urethra. Pessaries (devices placed inside the vagina in women) or surgery (e.g. suburethral sling) to elevate the urethra and/or bladder neck to increase the resistance to leak through the urethra are commonly used. Urethral bulking agents or pelvic muscle floor therapy are also employed to strengthen the closure pressure of the urethra in patients with stress UI. No pharmacologic agents are currently available to treat stress UI. For urge UI, medications or electrical stimulation aimed at relaxation of the detrusor muscle, including anticholinergics, are used. For overflow or obstructive UI, treatments are aimed at shrinking or removing the obstruction, such as medications to shrink the prostate, prostatectomy or mass removal. For neurogenic UI, surgery for diversion or implant placement may be utilized.

Sildenafil (Viagra) has been well studied and used extensively in males to treat erectile dysfunction. Phosphodiesterase 5 (PDE5) inhibitors, including sildenafil, are potent vasodilators that enhance tissue perfusion, relax smooth muscle of the vasculature and bladder, and stimulate skeletal muscle protein synthesis. It has been reported to improve lower urinary tract symptoms, including urge UI and benign prostatic hyperplasia (BPH) in men. In our team's recent study using sildenafil for treatment of UI in women, the investigators found improvement in quality of life and a decrease in the number of incontinence episodes in women taking sildenafil. Higher sildenafil plasma levels were associated with greater improvement in symptoms. While the types of UI in women are somewhat different than in men, studies have shown improvements in UI in both sexes.

Thus, the investigators propose to conduct a two month randomized, placebo-controlled crossover trial of sildenafil in male and female adult SCI patients with UI to assess the therapeutic potential of sildenafil to reduce the symptoms of urinary leakage.

Aims:

Aim 1: To determine whether sildenafil will decrease episodes of leakage of UI in adult women and men with SCI.

Aim 2: To determine the effects of sildenafil on the subjective measures of UI, including quality of life.

Experimental Protocol:

Investigators will study patients with spinal cord injuries (aged 18-70) with current urine leakage of more than 3 times/week (n=24). Subjects will undergo a double blinded randomized cross over treatment of sildenafil (20mg TID) and placebo. Each treatment period will last 4 weeks with a 2 week washout between treatment periods.

Before and after each treatment period, subjects will undergo testing which will consist of measurements of urine post void residual volume (PVR), adverse event assessment, and questionnaires of quality of life and urinary health.

ELIGIBILITY:
Inclusion Criteria:

* Adults with spinal cord injury (SCI), 18-75 years of age, at the time of consent
* Have urinary incontinence (UI), with at least 3 leakage episodes/week
* Have urodynamics assessment on file with their provider in past 3 years. If no historical data on file, subject may complete prior to study visit 1.
* Willing and able to comply with study procedures
* Willing and able to provide written informed consent

Exclusion Criteria:

* In phone prescreen, delighted or pleased with current quality of life due to urinary symptoms.
* Indwelling catheter
* History of greater than 4 urinary tract infections per year
* Multiple sclerosis
* Significant heart, liver, kidney, pulmonary, blood, autoimmune or peripheral vascular disease
* Systolic blood pressure <90 or >170, diastolic blood pressure <50 or >110 after repeated evaluation with proper cuff. This range is the acceptable range stated in the prescribing information for sildenafil (>90/50 and <170/110)
* Active cancer
* HIV, Hepatitis B, or Hepatitis C
* Use of systemic nitrates, anabolic steroids, corticosteroids, or long acting PDE5 inhibitors in the past 1 month
* Use of short acting PDE5 inhibitors in the past 1 week
* Use of alpha blockers, anticholinergic agents, bethanechol, or other UI treatment within the past 2 weeks ( 3 weeks for long acting muscarinic receptor antagonists)
* Known allergic reaction to any agent under investigation or required by the protocol
* Females who are pregnant or lactating
* Atonic bladder or high detrusor and high pelvic floor muscle pressure based on previous cystometrogram (CMG) (on file with their provider) that would place subjects at risk for kidney injury
* Any medical condition that, in the opinion of the investigator, would place the subject at increased risk for participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Bladder Leakage as measured by 5 day bladder diary at Baseline | baseline
  Bladder leakage will be measured by bladder diary, which will be kept for five- 24 hours periods at baseline. Subjects will be asked to record the number of leaks each day. Data will be calculated by summing total number of leaks over the 5 day recording period and dividing the sum by 5, resulting in average leaks per day.
Bladder Leakage as measured by 5 day bladder diary after 4 weeks of Sildenafil Treatment | after 4 weeks of sildenafil treatment
  Bladder leakage will be measured by bladder diary, which will be kept for five 24 hours periods in the last week of the 4 weeks of sildenafil treatment.
Bladder Leakage as measured by 5 day bladder diary after 4 weeks of Placebo Treatment | after 4 weeks of placebo treatment
  Bladder leakage will be measured by bladder diary, which will be kept for five 24 hours periods in the last week of the 4 weeks of placebo treatment.

SECONDARY OUTCOMES:
Blood sildenafil levels as measured by Liquid Chromatography Mass Spectrometry (LCMS) at baseline | baseline
  Sildenafil levels will be measured in plasma samples taken at baseline using a Liquid Chromatography Mass Spectrometry-Mass Spectrometry (LCMS-MS) method. Data will be reported as ng/ml.
Blood sildenafil levels as measured by Liquid Chromatography Mass Spectrometry (LCMS) after 4 weeks of sildenafil treatment | after 4 weeks of sildenafil treatment
  Sildenafil levels will be measured in plasma samples taken after 4 weeks of sildenafil treatment using a Liquid Chromatography Mass Spectrometry-Mass Spectrometry (LCMS-MS) method. Data will be reported as ng/ml.
Blood sildenafil levels as measured by Liquid Chromatography Mass Spectrometry (LCMS) after 4 weeks of placebo treatment | after 4 weeks of placebo treatment
  Sildenafil levels will be measured in plasma samples taken after 4 weeks of placebo treatment using a Liquid Chromatography Mass Spectrometry-Mass Spectrometry (LCMS-MS) method. Data will be reported as ng/ml.
Post void residual urine volume as measured by ultrasound bladder scanner at baseline | baseline
  Post void residual urine volume is measured using an ultrasound bladder scanner. To perform this test, the research subject empties their bladder and then the bladder scanner is used to measure any remaining urine in the bladder. Results will be reported as mL urine remaining.
Post void residual urine volume as measured by ultrasound bladder scanner after 4 weeks of sildenafil treatment | after 4 weeks of sildenafil treatment
  Post void residual urine volume is measured using an ultrasound bladder scanner. To perform this test, the research subject empties their bladder and then the bladder scanner is used to measure any remaining urine in the bladder. Results will be reported as mL urine remaining.
Post void residual urine volume as measured by ultrasound bladder scanner after 4 weeks of placebo treatment | after 4 weeks of placebo treatment
  Post void residual urine volume is measured using an ultrasound bladder scanner. To perform this test, the research subject empties their bladder and then the bladder scanner is used to measure any remaining urine in the bladder. Results will be reported as mL urine remaining.
Urinary symptoms as measured by the American Urological Association Symptom Score at baseline | baseline
  Urinary symptoms will be assessed using the American Urological Association (AUA) Symptom Score, a 7 item questionnaire that assess how bothersome urinary problems are and if treatment is effective. The AUA symptom score yields one overall score (range 0 - 35, with higher scores indicating higher severity). Total scores of 0-7 mild symptoms; 8-19 moderate symptoms; 20-35 severe symptoms
Urinary symptoms as measured by the American Urological Association Symptom Score after 4 weeks of sildenafil treatment | after 4 weeks of sildenafil treatment
  Urinary symptoms will be assessed using the American Urological Association (AUA) Symptom Score, a 7 item questionnaire that assess how bothersome urinary problems are and if treatment is effective. The AUA symptom score yields one overall score (range 0 - 35, with higher scores indicating higher severity). Total scores of 0-7 mild symptoms; 8-19 moderate symptoms; 20-35 severe symptoms
Urinary symptoms as measured by the American Urological Association Symptom Score after 4 weeks of placebo treatment | after 4 weeks of placebo treatment
  Urinary symptoms will be assessed using the American Urological Association (AUA) Symptom Score, a 7 item questionnaire that assess how bothersome urinary problems are and if treatment is effective. The AUA symptom score yields one overall score (range 0 - 35, with higher scores indicating higher severity). Total scores of 0-7 mild symptoms; 8-19 moderate symptoms; 20-35 severe symptoms
Bladder dysfunction as measured by the Neurogenic Bladder Symptom Score at baseline | baseline
  The Neurogenic Bladder Symptom Score (NBSS) is a validated questionnaire that assess symptoms of bladder dysfunction due to spinal cord injury. Three distinct domains are assessed: incontinence; storage and voiding; and consequences. Scores can range from 0 (no symptoms at all) to 74 (maximum symptoms).
Bladder dysfunction as measured by the Neurogenic Bladder Symptom Score after 4 weeks of sildenafil treatment | after 4 weeks of sildenafil treatment
  The Neurogenic Bladder Symptom Score (NBSS) is a validated questionnaire that assess symptoms of bladder dysfunction due to spinal cord injury. Three distinct domains are assessed: incontinence; storage and voiding; and consequences. Scores can range from 0 (no symptoms at all) to 74 (maximum symptoms).
Bladder dysfunction as measured by the Neurogenic Bladder Symptom Score after 4 weeks of placebo treatment | after 4 weeks of placebo treatment
  The Neurogenic Bladder Symptom Score (NBSS) is a validated questionnaire that assess symptoms of bladder dysfunction due to spinal cord injury. Three distinct domains are assessed: incontinence; storage and voiding; and consequences. Scores can range from 0 (no symptoms at all) to 74 (maximum symptoms).
Perception of bladder conditions as measured by the Patient Perception of Bladder Symptoms questionnaire at baseline | baseline
  The Patient Perceived Bladder Condition (PPBC) is a one item assessment measuring the severity of bladder problems with a likert scale with a range from 1 (best) to 6 (worst).
Perception of bladder conditions as measured by the Patient Perception of Bladder Symptoms questionnaire after 4 weeks of sildenafil treatment | after 4 weeks of sildenafil treatment
  The Patient Perceived Bladder Condition (PPBC) is a one item assessment measuring the severity of bladder problems with a likert scale with a range from 1 (best) to 6 (worst).
Perception of bladder conditions as measured by the Patient Perception of Bladder Symptoms questionnaire after 4 weeks of placebo treatment | after 4 weeks of placebo treatment
  The Patient Perceived Bladder Condition (PPBC) is a one item assessment measuring the severity of bladder problems with a likert scale with a range from 1 (best) to 6 (worst).
Urinary Symptoms Interference as measured by Pelvic Floor Impact Questionnaire at baseline | baseline
  Pelvic Floor Impact Questionnaire (PFIQ-7) is a 7 item questionnaire measuring how much urinary symptoms affect activities of daily living, relationships and feelings. Each question is answered three times each, corresponding to the three scales - bladder/urine; bowel/rectum; vagina/penis). Responses for each question range from "not at all" (0) to "quite a bit" (3). Each scale is scored separately by calculating the mean of all seven questions and multiplying that number by 100 and then dividing by 3. Scale scores range from 0-100 with lower scores indicating less effect on quality of life. PFIQ-7 summary score is calculated by summing all three subscale scores (range 0-300).
Urinary Symptoms Interference as measured by Pelvic Floor Impact Questionnaire after 4 weeks of sildenafil treatment | after 4 weeks of sildenafil treatment
  Pelvic Floor Impact Questionnaire (PFIQ-7) is a 7 item questionnaire measuring how much urinary symptoms affect activities of daily living, relationships and feelings. Each question is answered three times each, corresponding to the three scales - bladder/urine; bowel/rectum; vagina/penis). Responses for each question range from "not at all" (0) to "quite a bit" (3). Each scale is scored separately by calculating the mean of all seven questions and multiplying that number by 100 and then dividing by 3. Scale scores range from 0-100 with lower scores indicating less effect on quality of life. PFIQ-7 summary score is calculated by summing all three subscale scores (range 0-300).
Urinary Symptoms Interference as measured by Pelvic Floor Impact Questionnaire after 4 weeks of placebo treatment | after 4 weeks of placebo treatment
  Pelvic Floor Impact Questionnaire (PFIQ-7) is a 7 item questionnaire measuring how much urinary symptoms affect activities of daily living, relationships and feelings. Each question is answered three times each, corresponding to the three scales - bladder/urine; bowel/rectum; vagina/penis). Responses for each question range from "not at all" (0) to "quite a bit" (3). Each scale is scored separately by calculating the mean of all seven questions and multiplying that number by 100 and then dividing by 3. Scale scores range from 0-100 with lower scores indicating less effect on quality of life. PFIQ-7 summary score is calculated by summing all three subscale scores (range 0-300).

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Vincent, MD, Principal Investigator — University of Texas
Locations (2):
- United States (2):
  - Texas A&M University, College Station, Texas
  - University of Texas Medical Branch, Galveston, Texas

IPD SHARING:
Plan to Share IPD: No